CLINICAL TRIAL: NCT02745431
Title: Oxytocin Effects on Likeability After Being Liked or Disliked
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-06
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-11

CONDITIONS: Social Behavior
Keywords: Likeability; Being liked
MeSH Terms: conditions — Social Behavior | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin nasal spray (Experimental): Oxytocin nasal spray
  Interventions: Drug: Oxytocin
- Placebo nasal spray (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin nasal spray
Drug: Placebo
  Arms: Placebo nasal spray

SUMMARY:
The current study aimed to investigate oxytocin effect on the response after the experience of being liked or disliked.

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo controlled design study, the researchers aimed to investigate the intranasal OXT (40IU) treatment on rating response after being liked or disliked in healthy male subjects. All subjects completed a range of questionnaires measuring personality and affective traits and levels of anxiety: Positive and Negative Affect Schedule (PANAS) , State-Trait Anxiety Inventory (STAI) , Beck Depression Inventory (BDI), Cheek and Buss shyness Scale (CBSS),Autism Spectrum Quotient (ASQ), Empathy Quotient(EQ) before self-administration.Study participants were led to believe that other participants had formed an opinion on their likability based on their appearance in a photograph and they passively viewed the responses (like or dislike) from 'other participants'. After that, they rated 'other participants' about likeability (how much do you like the person), accuracy (have you seen the person), feeling (how good do you feel), and tendency (how much would do like have him/her as a friend). Likeability, tendency, feeling and accuracy were included into analysis as dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorder

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Oxytocin effect on likeability after being liked or disliked | 2 hour
  Likeability rating was included into analysis as dependent factor.

SECONDARY OUTCOMES:
Relationship status may influence oxytocin effect | 2 hour
  subjects were subdivided into two subgroups

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao W, Ma X, Le J, Ling A, Xin F, Kou J, Zhang Y, Luo R, Becker B, Kendrick KM. Oxytocin biases men to be more or less tolerant of others' dislike dependent upon their relationship status. Psychoneuroendocrinology. 2018 Feb;88:167-172. doi: 10.1016/j.psyneuen.2017.12.010. Epub 2017 Dec 22. PMID 29304421